CLINICAL TRIAL: NCT03816033
Title: Multi-catheter Cryotherapy Versus Radiofrequency Catheter Ablation for the Treatment of Standard and Resistant Arrhythmias
Brief Title: Cryotherapy Versus Radiofrequency Catheter Ablation Research Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. George's Hospital, London (Other)
Responsible Party: Principal Investigator, Dr. Mark M. Gallagher, Consultant Cardiologist and electrophysiologist, St. George's Hospital, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS236684
Record Dates: First submitted 2018-11-06; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia; Wpw; Ventricular Tachycardia
Keywords: catheter ablation techniques
MeSH Terms: conditions — Atrial Fibrillation; Wolff-Parkinson-White Syndrome; Tachycardia, Ventricular | interventions — Cryotherapy; Catheter Ablation

STUDY DESIGN:
Intervention Model Description: This is a 1:1 randomised clinical controlled trial or a set of them, in our extensive program of research.
Who Masked: Outcomes Assessor
Masking Description: The physiologist analysing the Holter results and/or loop recorders for recurrence of arrhythmia will not know the randomised treatment for the study participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Active Comparator): Cryotherapy ablation energy will be utilised in the catheter ablation procedure
  Interventions: Procedure: Cryotherapy
- Radiofrequency (Active Comparator): Radiofrequency ablation energy will be utilised in the catheter ablation procedure
  Interventions: Procedure: radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Cryotherapy — Catheter ablation treatment for the treatment of the studied arrhythmias
  Arms: Cryotherapy
Procedure: radiofrequency catheter ablation — Catheter ablation treatment for the treatment of the studied arrhythmias
  Arms: Radiofrequency

SUMMARY:
A program of research has been set up at St. George's Hospital, London studyng the practicalities of catheter ablation. The current practice of catheter ablation is being studied for a range of arrhythmias including PAF, persistent AF, advanced persistent AF and resistant WPW.

DETAILED DESCRIPTION:
The study design will be a separate randomised clinical trial for each of the arrhythmias studied. There will be 1:1 randomisation to either the cryotherapy protocol or RF protocol. Arrhythmia patients already under the care of this cardiac centre, who have already opted for catheter ablation treatment will be approached to ask if they will also be willing to participate in this longterm research program.

The protocols for each different arrhythmia are in line with current practice and knowledge and utilising current technology. In the program, the investigators have 1 or 2 protocols that mildly differ from conventional use but have already passed through initial experience with publication on this- this is the multi-catheter cryocatheter approach.

Acute procedural outcomes, short, medium and longterm success will be recorded for each patient, in addition to patient or participant experience and quality of life outcomes.

The catheter ablation research program has passed through ethical panel review in London and has the potential to become a multi-centre study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients under the care of the Arrhythmia Service at St. George's Hospital with one of the studied arrhythmia (PAF, persistent AF etc), awaiting catheter ablation treatment will be eligible for inclusion to the program of research

Exclusion Criteria:

* Vulnerable patients will be excluded- e.g. active cancer, inability to consent
* Paediatric patients will not be studied
* Patients awaiting standard SVT catheter ablation treatment

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence of the treated arrhythmia at 6 months | 6 months
  Recurrence of the treated arrhythmia or related tachycardia will be recorded in a single timeframe of 6 months. The method for recording recurrence will be from Holter or via loop recorder download.
Recurrence of the treated arrhythmia at 12 months | 12 months
  Recurrence of the treated arrhythmia or related tachycardia will be recorded in a single timeframe of 12 months. The method for recording recurrence will be from Holter or via loop recorder download.
Recurrence of the treated arrhythmia at 24 months | 24 months
  Recurrence of the treated arrhythmia or related tachycardia will be recorded in a single timeframe of 24 months. The method for recording recurrence will be from Holter or via loop recorder download.

SECONDARY OUTCOMES:
The rate of major adverse cerebrovascular and/or cardiovascular complications (defined as MI, CVA, vascular, oesophageal trauma, phrenic nerve injury) will be recorded | 24 months
  A record of MACCE (MI, CVA, vascular, oesophageal trauma, phrenic nerve injury) will be recorded for all participants for 24 months
To record the patient quality of life improvement by filling in a Short Form-36 questionnaire | 24 months
  The validated questionnaire is called the General Health Short Form-36 questionnaire. It is a general health questionnaire with 36 questions. The scoring system works from 0-100. The higher the score, the more favourable the general well-being of the patient or participant.

CONTACTS AND LOCATIONS:
Locations (1):
- St.George's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The research data will be kep in a closed system within our NHS centre to the direct care team and researchers. Once anonymised data is available to be presented, it will be presented on an international stage and publications are expected, in respected journals.

REFERENCES:
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Ciconte G, Ottaviano L, de Asmundis C, Baltogiannis G, Conte G, Sieira J, Di Giovanni G, Saitoh Y, Irfan G, Mugnai G, Storti C, Montenero AS, Chierchia GB, Brugada P. Pulmonary vein isolation as index procedure for persistent atrial fibrillation: One-year clinical outcome after ablation using the second-generation cryoballoon. Heart Rhythm. 2015 Jan;12(1):60-6. doi: 10.1016/j.hrthm.2014.09.063. Epub 2014 Oct 2. PMID 25281891
- [Background] Hunter RJ, Baker V, Finlay MC, Duncan ER, Lovell MJ, Tayebjee MH, Ullah W, Siddiqui MS, McLEAN A, Richmond L, Kirkby C, Ginks MR, Dhinoja M, Sporton S, Earley MJ, Schilling RJ. Point-by-Point Radiofrequency Ablation Versus the Cryoballoon or a Novel Combined Approach: A Randomized Trial Comparing 3 Methods of Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation (The Cryo Versus RF Trial). J Cardiovasc Electrophysiol. 2015 Dec;26(12):1307-14. doi: 10.1111/jce.12846. Epub 2015 Nov 25. PMID 26727045
- [Background] Bisleri G, Rosati F, Bontempi L, Curnis A, Muneretto C. Hybrid approach for the treatment of long-standing persistent atrial fibrillation: electrophysiological findings and clinical results. Eur J Cardiothorac Surg. 2013 Nov;44(5):919-23. doi: 10.1093/ejcts/ezt115. Epub 2013 Mar 8. PMID 23475587
- [Background] Haissaguerre M, Hocini M, Sanders P, Takahashi Y, Rotter M, Sacher F, Rostock T, Hsu LF, Jonsson A, O'Neill MD, Bordachar P, Reuter S, Roudaut R, Clementy J, Jais P. Localized sources maintaining atrial fibrillation organized by prior ablation. Circulation. 2006 Feb 7;113(5):616-25. doi: 10.1161/CIRCULATIONAHA.105.546648. PMID 16461833
- [Background] Tada H, Yamada M, Naito S, Nogami A, Oshima S, Taniguchi K. Radiofrequency catheter ablation within the coronary sinus eliminates a macro-reentrant atrial tachycardia: importance of mapping in the coronary sinus. J Interv Card Electrophysiol. 2006 Jan;15(1):35-41. doi: 10.1007/s10840-006-6310-2. PMID 16680548
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, Della Bella P, Hindricks G, Jais P, Josephson ME, Kautzner J, Kay GN, Kuck KH, Lerman BB, Marchlinski F, Reddy V, Schalij MJ, Schilling R, Soejima K, Wilber D; European Heart Rhythm Association (EHRA); Registered Branch of the European Society of Cardiology (ESC); Heart Rhythm Society (HRS); American College of Cardiology (ACC); American Heart Association (AHA). EHRA/HRS Expert Consensus on Catheter Ablation of Ventricular Arrhythmias: developed in a partnership with the European Heart Rhythm Association (EHRA), a Registered Branch of the European Society of Cardiology (ESC), and the Heart Rhythm Society (HRS); in collaboration with the American College of Cardiology (ACC) and the American Heart Association (AHA). Heart Rhythm. 2009 Jun;6(6):886-933. doi: 10.1016/j.hrthm.2009.04.030. No abstract available. PMID 19467519
- [Background] Andrade JG, Dubuc M, Guerra PG, Macle L, Mondesert B, Rivard L, Roy D, Talajic M, Thibault B, Khairy P. The biophysics and biomechanics of cryoballoon ablation. Pacing Clin Electrophysiol. 2012 Sep;35(9):1162-8. doi: 10.1111/j.1540-8159.2012.03436.x. Epub 2012 Jun 5. PMID 22671922